CLINICAL TRIAL: NCT05086627
Title: A Single -Centers, Randomized, Open-label, Controlled Phase Ⅱ Clinical Trial of Short-course Radiotherapy Followed by Tislelizumab + CapeOX in the Treatment for Locally Advanced Rectal Cancer
Brief Title: Short-course Radiotherapy Followed by Tislelizumab + CapeOX in the Treatment for Locally Advanced Rectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hebei Medical University Fourth Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021104
Record Dates: First submitted 2021-09-15; First posted 2021-10-21 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Locally Advanced Rectal Cancer
Keywords: Locally advanced rectal cancer; Neoadjuvant radiotherapy; Immune checkpoint inhibitors; Programmed death-1 inhibitor
MeSH Terms: interventions — tislelizumab; XELOX

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Short-course radiotherapy sequential Tislelizumab combined with CapeOX (group A) (Experimental): Standard SCRT: A total radiation dose of 25 Gy was delivered in 5 fractions (from day 1 to 5)
  Sequential treatment period: After resting for 3-7 days following completion of SCRT, patients were treated with 4 cycles of CapeOX (Oxaliplatin 130 mg/m2 intravenously, day 1; Capecitabine 1000 mg/m2, Bid,days 1-14) and an additional intravenous infusion of 200mg Tislelizumab on the first day of each cycle of CapeOX.
  Surgery: After 3 weeks of the completion of neoadjuvant therapy, the TME surgery was performed.
  Postoperative adjuvant chemotherapy: Whether postoperative chemotherapy was implemented mainly depended on the patient's wishes, and 2 cycles of CapeOX with or without Tislelizumab will be undergone to these willing cases.
  Interventions: Drug: Tislelizumab; Radiation: Short-course radiotherapy; Drug: Capecitabine+Oxaliplatin
- Short-course radiotherapy sequential CapeOX (group B) (Active Comparator): Standard SCRT: A total radiation dose of 25 Gy was delivered in 5 fractions (from day 1 to 5)
  Sequential treatment period: After resting for 3-7 days following completion of SCRT, patients were treated with 4 cycles of CapeOX (Oxaliplatin 130 mg/m2 intravenously, day 1; Capecitabine 1000 mg/m2, Bid,days 1-14).
  Surgery: After 3 weeks of the completion of neoadjuvant therapy, the TME surgery was performed.
  Postoperative adjuvant chemotherapy: Whether postoperative chemotherapy was implemented mainly depended on the patient's wishes, and 2 cycles of CapeOX will be undergone to these willing cases.
  Interventions: Radiation: Short-course radiotherapy; Drug: Capecitabine+Oxaliplatin

INTERVENTIONS:
Drug: Tislelizumab — Patients were treated with Tislelizumab on the first day of each cycle of CapeOX (Capecitabine+Oxaliplatin).
  Arms: Short-course radiotherapy sequential Tislelizumab combined with CapeOX (group A)
Radiation: Short-course radiotherapy — Patients were treated with short-course neoadjuvant radiotherapy
Drug: Capecitabine+Oxaliplatin — Patients were treated with neoadjuvant chemotherapy with CapeOX (Capecitabine+Oxaliplatin).

SUMMARY:
This study is a single-center, prospective, open-label, randomized controlled clinical study, and the purpose of this study was to compare the pathological complete response rate (PCR) of patients with locally advanced rectal cancer treated with short-course radiotherapy sequential Tislelizumab combined with CapeOX (group A) versus short-course radiotherapy sequential CapeOX (group B). A total of 100 patients with locally advanced rectal cancer will be enrolled in the study. These patients were randomly assigned to the experimental group (group A) and the control group (group B) in a ratio of 1:1.

DETAILED DESCRIPTION:
Baseline examnation: All enrolled patients in this study, in addition to routine laboratory and imaging examinations such as blood routine, blood biochemistry, serum tumor markers (Incl. CEA, CA-199, CA-724 β2-microglobulin, Ferroprotein), chest CT, abdominal and pelvic MRI, etc., were required to undergo KRAS, NRAS, BREF, PD-L1, MMR/MSS testings before SCRT, and blood lymphocyte subgroups were analyzed before SCRT, systemic therapy, and surgery.

Subjects in group A will be treated according to the following treatment plan:

Standard SCRT: A total radiation dose of 25 Gy was delivered in 5 fractions (from day 1 to 5)

Sequential treatment period: After resting for 3-7 days following completion of SCRT, patients were treated with 4 cycles of CapeOX (Oxaliplatin 130 mg/m2 intravenously, day 1; Capecitabine 1000 mg/m2, Bid,days 1-14) and an additional intravenous infusion of 200mg Tislelizumab on the first day of each cycle of CapeOX.

Surgery: After 3 weeks of the completion of neoadjuvant therapy, the TME surgery was performed.

Postoperative adjuvant chemotherapy:Whether postoperative chemotherapy was implemented mainly depended on the patient's wishes, and 2 cycles of CapeOX with or without Tislelizumab will be undergone to these willing cases.

Subjects in group B will be treated according to the following treatment plan:

Standard SCRT: A total radiation dose of 25 Gy was delivered in 5 fractions (from day 1 to 5)

Sequential treatment period: After resting for 3-7 days following completion of SCRT, patients were treated with 4 cycles of CapeOX (Oxaliplatin 130 mg/m2 intravenously, day 1; Capecitabine 1000 mg/m2, Bid,days 1-14).

Surgery: After 3 weeks of the completion of neoadjuvant therapy, the TME surgery was performed.

Postoperative adjuvant chemotherapy:Whether postoperative chemotherapy was implemented mainly depended on the patient's wishes, and 2 cycles of CapeOX will be undergone to these willing cases.

Endpoint: The primary endpoint was pCR rate. Secondary endpoints included MPR (TRG0+TRG1), 3-year PFS, 3-year OS, and treatment safety.

Follow-up records during treatment: For the duration of operation, the time required to complete the TME surgery and the amount of blood loss were recorded, and the impact of neoadjuvant therapy on the operation was observed. During the SCRT process, and the period of resting after SCRT, of the entire preoperative systemic treatment, of the resting after TME surgery, of the postoperative chemotherapy (these willing cases), the occurrence of adverse events (AE) of participants were closely monitored and actively responded.

ELIGIBILITY:
Inclusion Criteria:

Patients or their family members agree to participate in the study and sign the informed consent form;

Patients ≥ 18 and ≤75 years old, male or female;

ECOG performance status of 0 or 1;

Patients with histologically confirmed rectal adenocarcinoma;

The clinical diagnosis of chest CT, abdominal and pelvic enhanced MRI was T1-2N+M0 and cT3-4NanyM0 (the T and N stage was based on pelvic enhanced MRI+DWI, M stage was determined by liver enhanced MRI+DWI and chest CT, and if necessary, PET-CT was used);

The distance between the lower edge of the tumor and the anal edge is less than or equal to 10 cm;

No history of immune system diseases;

No history of immunodeficiency, including HIV positive;

No history of other malignancies;

No history of myocarditis;

No history of severe cardiovascular and cerebrovascular diseases;

No history of thyroid dysfunction;

No history of liver and kidney diseases;

No history of mental illness, no history of Infectious diseases;

No history of organ transplantation or allogeneic bone marrow transplantation;

There is no history of other systemic diseases other than the above diseases;

Voluntarily accept the neoadjuvant treatment scheme of radiotherapy, sequential chemotherapy / chemotherapy combined with immunotherapy;

Swallowing pills normally;

Rectal cancer without radiotherapy, chemotherapy, surgery, Chinese medicine anti-tumor treatment, etc.;

Surgical treatment is planned after neoadjuvant treatment.

Exclusion Criteria:

Patients who do not meet the above inclusion criteria;

Documented history of allergy to study drugs, including any component of Tislelizumab, capecitabine, oxaliplatin and other platinum drugs;

Patients who need to be treated with corticosteroid (dose equivalent to prednisone of >10 mg/day) or other immunosuppressive agents within 2 weeks prior to study drug administration; Major surgery or severe trauma within 4 weeks before the first use of the study drug;

Severe infection (CTCAE > 2) occurred within 4 weeks before the first use of the study drug; Baseline chest imaging revealed active pulmonary inflammation, signs and symptoms of infection within 14 days prior to the first use of the study drug, or oral or intravenous antibiotic therapy, except for prophylactic use of antibiotics;

Female patients who is pregnant or breastfeeding;

Patients who refuse to sign informed consent by themselves or their authorized persons;

Patients with poor cognitive ability, unable to answer questions, unable to fill in questionnaires or mental disorders;

Patients considered unsuitable for the study by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-08-20 (Actual)

PRIMARY OUTCOMES:
Pathological complete response rate | 1 week after surgery
  Pathological complete response rate was defined as the absence of viable tumour cells in the resected primary tumour specimen and all sampled regional lymph nodes (ypT0N0)

SECONDARY OUTCOMES:
major pathologic response (TRG0+TRG1) | 1 week after surgery
  TRG 0 indicates no remaining viable cancer cells (complete response); TRG 1 indicates a single cell or small groups of cancer cells (moderate response)
3-year PFS | 3 years from randomization
  PFS refers to the time from randomization to tumor progresses or death from any cause
3-year OS | 3 years from randomization
  OS refers to the time from randomization to death from any cause
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | through study completion, an average of 1 year
  Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] during treatment, including chemoradiotherapy, immunology, sugery

CONTACTS AND LOCATIONS:
Locations (1):
- Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei, China

IPD SHARING:
Plan to Share IPD: No